CLINICAL TRIAL: NCT06993584
Title: Pharmacokinetic Modelling of Levosimendan in Adults in Cardiogenic Shock With or Without Extracorporeal Membrane Oxygenation Support
Brief Title: Pharmacokinetic Modelling of Levosimendan in Adults
Acronym: MILADECMO
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Collaborators: University Hospital, Lille (Other); Amiens University Hospital, France (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2022/0346/HP; 2025-A00556-43 (Other: ANSM)
Record Dates: First submitted 2025-05-19; First posted 2025-05-29 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-04

CONDITIONS: Cardiogenic Shock
Keywords: cardiogenic shock; levosimendan; pharmacokinetics; ECMO; extracorporeal membrane oxygenation; ECLS
MeSH Terms: conditions — Shock, Cardiogenic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Months
Biospecimen Retention: Samples Without DNA — 1 aliquot of the 2 mL EDTA blood tube and 1 aliquot of the 4 mL heparinised tube
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Adult patients in cardiogenic shock — evaluate the elimination clearance of levosimendan (LVSMD) in the group without extracorporeal membrane oxygenation (ECMO) and in the group with ECMO.

SUMMARY:
In the light of current knowledge of the PK of levosimendan and its use in ECMO weaning, deciphering the mechanisms of inter-individual variability in exposure and response to levosimendan appears essential in order to better stratify patients eligible or not for this therapy and to adapt the treatment of patients in cardiogenic shock, with or without ECMO support, accordingly. The aim of this project is to use an innovative pharmacokinetic modelling approach based on clinico-biological data to study the key factors that could contribute to treatment failure in cardiogenic shock and to integrate them quantitatively for dose individualisation. The aim of this project is to conduct a prospective, multicentre, observational, comparative analysis, with minimal risks and constraints, to determine the concentrations of levosimendan and its metabolites during patient management in order to develop a pharmacokinetic model.

DETAILED DESCRIPTION:
Cardiogenic shock is a pathological condition characterised by cardiac failure inducing tissue hypoxia and organ hypoperfusion, which can lead to multiple organ failure and death. Extracorporeal membrane oxygenation (ECMO) is a circulatory support technique commonly used in the treatment of cardiogenic shock. This device reduces mortality in patients with refractory shock, i.e. those who do not respond, or only partially respond, to medical treatment including inotropic and vasopressor pharmacological support. ECMO is associated with significant pharmacokinetic (PK) changes related to volume of distribution (Vd) and clearance (CL), which may alter the efficacy of treatments. From a PK point of view, the addition of an extracorporeal circuit capable of sequestering and/or degrading drugs represents a challenge for dose adjustment. Levosimendan (LVSMD) is a drug authorised for the treatment of acute decompensated heart failure. It's a lipophilic drug (logP=2.16) and highly protein-bound (>97%), two properties that favour its sequestration in the ECMO circuit [2]. This hypothesis is reinforced by the recent publication of a RIPH3 study evaluating the PK of levosimendan in neonates and children in intensive care, whether or not assisted by ECMO (NCT03681379, Bourgoin P, Duflot T, Clin Pharmacokinet). The rationale for this project is based on the following hypotheses: 1°) Beneficial effects on renal function, pulmonary congestion, physical capacity and cardiac output have been observed with levosimendan in the management of cardiogenic shock [4] 2°) The use of antibiotics could alter the metabolism of LVSMD leading to a defect in the synthesis of the active metabolite. 3°) LVSMD is beneficial during weaning from ECMO and the contradictions in previously published results [5] could be attributed to a reduced half-life of the drug and/or OR-1896 due to adsorption phenomena on the ECMO circuit making the treatment less effective.

ELIGIBILITY:
Inclusion Criteria:

* Patient between 18 and 75 years of age admitted to an intensive care unit,
* Weight ≥ 50 kg,
* Patient with cardiogenic shock defined by a SCAI stage C, D, or E score.
* The medical team plans to initiate LVSMD treatment as part of the management of cardiogenic shock, according to the recommendations in the Summary of Product Characteristics (SmPC),
* Expected life expectancy > 48 hours,
* Patient affiliated with a social security scheme,
* Due to the life-threatening nature of cardiogenic shock, the patient or, where applicable, family members or trusted person are informed as soon as possible and their consent is requested for the possible continuation of this research. They may also object to the use of the patient's data (and blood samples) for this research.

Exclusion Criteria:

* Pregnant, childbearing, or breastfeeding women,
* Persons deprived of their liberty by an administrative or judicial decision, or persons placed under judicial protection/guardianship or curatorship.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with Lévosimendan (LVSMD) as part of their usual care for cardiogenic shock (60 with extracorporeal membrane oxygenation (ECMO) and 40 without ECMO)
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2027-07-30 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Elimination Clearance of Levosimendan (LVSMD) in Adult Patients in Cardiogenic Shock with Extracorporeal Membrane Oxygenation (ECMO) | At enrollment visit, hour 1, 2 and 6 and at hour 24, 26 and 32 after enrollment visit
  The clearance (CL) of Lévosimendan (LVSMD) will be determined by the ratio of the total dose administered to the exposure characterised by the area under the curve (AUC) over time (CL=Dose/AUC). In order to obtain an accurate estimate of the AUC, blood samples will be taken from a catheter already in place for the patient's therapeutic needs and will be taken at 0, 2, 6, 24, 26 and 32 hours after the start of an intravenous infusion of LVSMD at the dosage defined according to the recommendations in the Summary of Product Characteristics (SmPC).

SECONDARY OUTCOMES:
Success rate of weaning in the ECMO patient group | Hour 72 after enrollment visit
  The success rate in the extracorporeal membrane oxygenation (ECMO) group will be assessed by the proportion of patients weaned from ECMO within 72 hours of the end of the levosimendan (LVSMD) infusion. ECMO weanability is assessed according to the Extracorporeal Life Support Organization (ELSO) guidelines by a weaning test, initiated after myocardial recovery, defined by a reduction in amine requirements to a minimum threshold to achieve a mean arterial pressure (MAP) > 65 mmHg with an ECMO flow rate less than 2.5 L/min, usually performed for ECMO weaning. The weaning test is performed under an ECMO flow rate of 1L/min for 3 to 5 minutes, and is a success if the following parameters are obtained under low doses of amines: subaortic ITV > 12 cm/s, LVEF > 25-30%, absence of right ventricular dysfunction, central venous pressure < 10 mmHg and MAP > 60 mmHg
Hemodynamic success rate in the group without extracorporeal membrane oxygenation (ECMO) | Hour 72 after enrollment visit
  he success rate in the group without extracorporeal membrane oxygenation (ECMO) will be assessed by the proportion of patients with an increase in cardiac index of at least 20% associated with venous oxygen saturation > 65% within 72 hours following the end of the levosimendan (LVSMD) infusion, and/or improvement in hemodynamics (normalization of SvO2 and cardiac index > 2.2 L/min/m2 without increase or introduction of dobutamine).
Population-based pharmacokinetic model of LVSMD and its metabolites | Hours 48, 72, 96, 120, 144, 168, 336 and 504 after enrollment visit
  The population-based PK model, based on the results of the pediatric population study, will use a two-compartment model with first-order elimination for Lévosimendan (LVSMD). The appearance of metabolites will be modeled by transit compartments and their elimination will follow first-order kinetics. The collected clinical-biological data will be evaluated as covariates or as regressors (for time-dependent variables). Pharmacokinetic parameters will be evaluated according to a lognormal distribution (solutions > 0) and regressors according to a normal distribution. Pharmacokinetic parameters will be calculated in a global structural population model and individual parameters will be determined by Bayesian estimation. The final model will then be used to perform simulations to establish the dosage allowing similar exposure between patients supported by extracorporeal membrane oxygenation (ECMO) and patients without extracorporeal membrane oxygenation (ECMO) during cardiogenic shock.
Influence of a change in intestinal microbiota on the conversion of levosimendan into its active metabolite | Two rectal swabs 24 hours apart, one at enrollment visit and one at hour 24 after enrollment visit
  Given the metabolism of levosimendan to OR1896 by intestinal microbiota described in numerous studies, it seems legitimate to wonder whether inter-individual variability in response to treatment might not be linked to individual changes in intestinal microbiota. The aim is therefore to characterize the intestinal microbiota by swabbing and bioinformatic analysis, and to determine whether there are responder or non-responder profiles.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas TD DUFLOT, PharmD, Study Chair — pharmacology department, University Hospital of Rouen; Emmanuel BESNIER, MD, PHD, Study Chair — anesthesiology, University Hospital of Rouen
Locations (3):
- France (3):
  - Cardio-Thoracic-Vascular Resuscitation Department, university Hospital of Amiens, Amiens
  - Anesthesia Clinic - Resuscitation, University Hospital of Lile, Lille
  - Anesthesia-Resuscitation Department, University Rouen Hospital, Rouen

IPD SHARING:
Plan to Share IPD: No
The data provided will be the property of the sponsor and will be used solely for its own research activities.